CLINICAL TRIAL: NCT03524209
Title: Comparison of Thoracolumbar Back Pain After Brace Treatment Versus Percutaneous Instrumentation in Adult Pyogenic Spondylodiscitis Combined With Antibiotic Treatment
Brief Title: CORset Versus OstéoSynthese in Adult Pyogenic Spondylodiscitis
Acronym: COROSIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6751
Record Dates: First submitted 2018-03-12; First posted 2018-05-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Spondylodiscitis
Keywords: Spondylodiscitis; spinal infection; back pain; quality of life; fusion; minimal invasive surgery; brace treatment
MeSH Terms: conditions — Discitis; Back Pain | interventions — Braces

STUDY DESIGN:
Intervention Model Description: A prospective selection of patients with pyogenic spondylitis fulfilling above mentioned inclusion criteria is performed with subsequent randomization into treatment group 1 versus treatment group 2 after informed consent. Group1 are patients treated by minimally invasive surgery and group 2 are patients treated by thoracolumbar brace.
  Radiologic deformity assessment is performed on lateral thoracolumbar radiographs in standing position. A modified sagittal index measuring the angulation between cranial endplate of cranial vertebra and caudal endplate of the caudal vertebra as this parameter is normalized to 0°.
  Assessment of osteolysis at vertebral bodies on CT expressed as a ratio of vertebral body height in the mid-sagittal plane in comparison to non-infected vertebral bodies adjacent to the index level. Assessment of complete fusion, partial fusion, pseudarthrosis is performed on CT at 1-year FU.
  Type and length of antibiotic treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Other): Patients with spondylodiscitis are operated by percutaneous instrumentation and receive an antibiotic treatment according to the bacterium evidenced in the initial diagnostic intervertebral disc puncture (6 weeks to 3 months according to CRP course)
  Interventions: Device: Percutaneous instrumentation of the thoracolumbar spine
- Brace (Other): Patients with spondylodiscitis are wearing a thoracolumbar brace for 3 months and receive an antibiotic treatment according to the bacterium evidenced in the initial diagnostic intervertebral disc puncture (6 weeks to 3 months according to CRP course)
  Interventions: Other: Brace

INTERVENTIONS:
Device: Percutaneous instrumentation of the thoracolumbar spine — The spine is stabilized cranially and caudally of the level of spondylodiscitis. The percutaneous instrumentation consists of a rod and pedicle screw construct. The vertebrae are instrumented through minimal skin incisions using a fluoroscopic guidance or a spinal navigation system based on 3D imaging.
  Other Names: minimal invasive surgery (MIS)
  Arms: Surgery
Other: Brace — Brace treatment is associated in patients presenting back pain and a risk for vertebral body collapse due to infection with subsequent kyphotic deformity of the thoracolumbar spine
  Arms: Brace

SUMMARY:
Pyogenic spondylitis in adults is usually treated by antibiotics according to bacteria evidenced in a diagnostic intervertebral disc puncture. Brace treatment is associated in patients presenting back pain and a risk for vertebral body collapse due to infection with subsequent kyphotic deformity of the thoracolumbar spine. Percutaneous minimally invasive posterior spinal instrumentation has evolved over the last decade and indications in infections arouse over the last years. This procedure is interesting as it is performed through small skin incisions only. It avoids paravertebral muscle dissection and thus limits intraoperative bleeding and access morbidity. Recent retrospective data suggests that this internal fixation represents a theoretical advantage over brace treatment by lowering back pain and increasing patient's quality of life in the short run, up to 3 months, but no randomized study was published. The patient's autonomy, including walking ability and daily activities, might improve more rapidly after a percutaneous procedure. Additionally, the sagittal alignment of the thoracolumbar spine could be better maintained by internal fixation, which might prevent progression into kyphosis and improve long-term outcome. The hypothesis is the superiority of percutaneous minimally invasive instrumentation on brace treatment in term of quality of life, back pain and quality of osseous healing.

DETAILED DESCRIPTION:
Safety and efficacy of percutaneous for the indication of pyogenic spondylitis has been demonstrated retrospectively on small cohort studies, which is in line with our clinical experience. Although this therapeutic concept seems applicable to patients with spondylitis, the theoretical clinical benefit of minimally invasive surgery remains hypothetic and unclear compared to brace treatment, which might still be regarded as the gold standard.

ELIGIBILITY:
Inclusion criteria:

* adult patients presenting acute pyogenic spondylitis of the thoracolumbar spine
* back pain at a minimum of 4 out of 10 on VAS
* Diagnostic MRI and disc puncture + microbiological analysis required for antibiotic treatment and/or blood culture
* Vertebral body involvement (osteolysis) < 50% of VB height documented on CT

Exclusion criteria:

* postoperative pyogenic spondylitis or infection after spinal instrumentation spinal tuberculosis and mycosis
* contra-indications for surgery or general anaesthesia
* general septic conditions acute endocarditis documented by sonography
* patients presenting another major abcess or an epidural abscess
* Absence of vertebral body involvement (osteolysis) on CT or minor VB involvement less than 10% of VB height (surgery not indicated)
* Major destruction of vertebral body (>50%) on CT (surgery mandatory) Patients with concomitant bacterial endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Pre treatment
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Post treatment day 5
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Post treatment 6 weeks
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Post treatment 3 months
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Post treatment 6 months
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Post treatment 1 year
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)
Comparison of VAS for back pain for brace versus percutaneous instrumentation | Post treatment 2 years
  VAS score from 0 to 10 filled out by patients for clinical evaluation of primary outcome measure (pain)

SECONDARY OUTCOMES:
Comparison of quality of life (QoL) by EQ-5D for brace versus percutaneous instrumentation | Change of score between pre treatment and during 2 years after treatment
  EQ-5D-3L questionnaire filled out by the patients
- Comparison of influence of both treatment on kyphotic deformity - Comparison of fusion rates versus pseudarthrosis for both treatments | Change of measures between pre treatment and during 2 years after treatment
  Radiographic measurements by modified sagittal index on lateral radiographs in standing position
Analysis of correlation between kyhphosis / fusion and VAS / QoL scores | Change of measures between pre treatment and during 2 years after treatment
  Radiographic measurements by modified sagittal index on lateral radiographs in standing position
Course of CRP | Change of value between pre treatment and during 3 months after treatment
  Routine blood tests for documentation of CRP
Documentation of secondary complications after percutaneous instrumentation | Change between pre treatment and during 2 years after treatment
  Comparison of influence of both treatment

OTHER OUTCOMES:
Documentation, reporting and analysis of potential complications | Change between pre treatment and during 2 years after treatment
  Comparison of influence of both treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yann Philippe CHARLES, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg - Service de chirurgie du rachis
Locations (15):
- France (15):
  - CHU de Bordeaux - Hôpital Pellegrin - Unité d'orthopédie-traumatologie rachis I, Bordeaux
  - CHU de CAEN, Caen
  - Hôpital Beaujon - Service de Chirurgie Orthopédique et Traumatologie, Clichy
  - CHU François Mitterand - Bocage central - Service de Neurochirurgie, Dijon
  - CHU de GRENOBLE, Grenoble
  - CHU Lyon - Hôpital Pierre Wertheimer - Service de Neurochirurgie C et chirurgie du rachis, Lyon
  - CHU Marseille - Hôpital Timone - Service de chirurgie orthopédique et traumatologique, Marseille
  - Hôpital Gui de Chauliac - Service de Neurochirurgie, Montpellier
  - Hôpital Central - Service de Neurochirurgie, Nancy
  - CHU Hôtel Dieu - Service de Neurotraumatologie, Nantes
  - CHU Nice - Hôpital Pasteur 2 - Unité de Chirurgie Rachidienne, Nice
  - Hôpital Pitié - Salpêtrière - Service de Chirurgie orthopédique, Paris
  - Hôpital européen Georges-Pompidou - Service d'Orthopédie/Traumotologie, Paris
  - CHU Reims - Hôpital Maison Blanche - Service de Neurochirurgie, Reims
  - Hôpitaux Universitaires de Strasbourg - Service de chirurgie du rachis, Strasbourg

IPD SHARING:
Plan to Share IPD: No